CLINICAL TRIAL: NCT00773474
Title: A Phase II Study of Lonafarnib in Patients With Metastatic Breast Cancer
Brief Title: Lonafarnib in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding terminated
Sponsor: George Sledge (Other)
Collaborators: Schering-Plough (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, George Sledge, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG BRE07-126
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lonafarnib (Experimental): All registered patients will be treated with Lonafarnib 200 mg PO BID daily on days 1-21 of every 21-day cycle until progression of disease, unacceptable toxicity, or investigator's discretion.
  Interventions: Drug: Lonafarnib

INTERVENTIONS:
Drug: Lonafarnib — All registered patients will be treated with Lonafarnib 200 mg PO BID daily on days 1-21 of every 21-day cycle until progression of disease, unacceptable toxicity, or investigator's discretion.

SUMMARY:
A published phase 2 study reported that lonafarnib was administered as a single agent via continuous or intermittent oral dosing to 76 women with advanced breast cancer who were previously treated with chemotherapy and/or with endocrine therapy. Objective response rates of approximately 10% were observed. This study will determine the rate of progression-free survival of patients with metastatic breast cancer who receive lonafarnib.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study

Patients will be treated with lonafarnib 200 mg PO BID daily on days 1-21 of every 21-day cycle until progression of disease, unacceptable toxicity, or investigator's discretion.

1 Cycle = 21 days of lonafarnib (plus the time required to recover from toxicity if encountered).

ECOG Performance Status 0-1

Life Expectancy: Not Specified

Hematopoietic:

* Platelets > 100 K/mm3
* Absolute Neutrophil Count (ANC) > 1.2 K/mm3
* Hemoglobin ≥ 9 g/dl
* Serum potassium ≥ 3.3 mmol/L

Hepatic:

* Aspartate transaminase (AST) ≤ 5.0 x ULN
* Alanine transaminase (ALT) ≤ 5.0 x ULN
* Total bilirubin < 1.5 x ULN

Renal:

* Calculated creatinine clearance (using Cockcroft-Gault formula) > 45 cc/min

Cardiovascular:

* No history of Torsades de Pointes, ventricular tachycardia, ventricular fibrillation or ventricular flutter

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed adenocarcinoma of the breast with locally advanced or metastatic disease.
* Must be able and willing to enroll in the companion study entitled "Predicting Response and Toxicity in Patients Receiving Lonafarnib for Breast Cancer: A Multicenter Genomic, Proteomic and Pharmacogenomic Correlative Study: Hoosier Oncology Group COE-03."
* Must have measurable disease per RECIST as evaluated by imaging within 28 days prior to registration for protocol therapy.
* Must be willing to not drink grapefruit juice for the duration of lonafarnib therapy.
* Previously radiated area(s) must not be the only site of disease for study entry.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time of consent until at least 90 days following completion of study treatment.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to registration for protocol therapy. Subjects are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Females must not be breastfeeding.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years

Exclusion Criteria:

* No history or radiologic evidence of CNS metastases including previously treated, resected or asymptomatic brain lesions or leptomeningeal involvement (head CT or MRI must be obtained within 42 days prior to registration for protocol therapy).
* No treatment with any investigational agent within 30 days prior to registration for protocol therapy.
* No history of Torsades de Pointes, ventricular tachycardia, ventricular fibrillation or ventricular flutter.
* No history of syncope.
* No history of seizures.
* No prolonged QTc interval > 450msec on pre-entry electrocardiogram obtained within 28 days prior to registration for protocol therapy.
* No history of hypokalemia that cannot be corrected prior to registration for protocol therapy.
* No radiation within 14 days prior to registration for protocol therapy. Patients must have recovered from the acute toxic effects prior to registration for protocol therapy.
* No prior chemotherapy within 21 days prior to registration for protocol therapy.
* No clinically active serious infections as judged by the treating investigator (CTC v3, > Grade 2) including known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Following concomitant medications must be discontinued 7 days prior to registration for protocol therapy and for the duration of lonafarnib therapy: bisphosphonates, including but not limited to etidronate (Didronel), pamidronate (Aredia), alendronate (Fosamax), risedronate (Actonel), zoledronate (Zometa or Reclast), ibandronate (Boniva), ethinylestradiol, gestodene, itraconazole, ketoconazole, cimetidine, erythromycin, carbamazepine, high dose chronic steroids, phenobarbital, phenytoin, rifampin (rifampicin), sulfinpyrazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Sledge, M.D., Principal Investigator — Hoosier Cancer Research Network; Brian Leland-Jones, M.D., Principal Investigator — Hoosier Cancer Research Network
Locations (6):
- United States (6):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Ireland Cancer Center - University Hospitals of Cleveland, Cleveland, Ohio

REFERENCES:
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lonafarnib
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lonafarnib
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 56 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Primary Tumor Diagnosis [Number; unit: participants] — Participants can have more than one primary tumor diagnosis. The sum of all tumor diagnoses can/will be greater than the number of participants.
  participants
    Breast Carcinoma | 14
    Ductal Breast Carcinoma | 20
    Lobular Breast Carcinoma | 1
    Other | 1
Estrogen Receptor (ER)/Progesterone Receptor (PR)/ HER2 Status [Number; unit: participants] — Hormone Receptor Status. Each participant can have 0-3 possible HR statuses, consequently the sum of all HR statuses will be greater than the number of participants.
  participants
    ER- | 9
    ER+ | 15
    PR- | 13
    PR+ | 11
    HER2- | 17
    HER2+ | 3
    Unknown | 4
Number of Prior Therapies [Median (Full Range); unit: Prior Therapies] | 8.4 [0 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To determine progression-free survival of lonafarnib in patients with metastatic breast cancer.
Time Frame: 18 months
Population: 20 participants were eligible for analysis via the Kaplan-Meier method. PFS assessed via RECIST criteria.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Lonafarnib
Number analyzed (Participants) | 20
days | 65.5 [60 to 125]

2. Secondary Outcome: Overall Response Rate
Description: To determine overall response rate.
Time Frame: 18 months
Population: 17 participants were evaluable for Overall Response Rate analysis using RECIST criteria.
Measure: Number; unit: participants
Arm/Group | Lonafarnib
Number analyzed (Participants) | 17
participants
  CR | 0
  PR | 0
  SD | 5
  PD | 12

3. Secondary Outcome: Toxicity Profile of Lonafarib
Description: To determine the toxicity profile of lonafarnib in this patient population.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Lonafarnib
Number analyzed (Participants) | 29
participants
  Grade 3/4 Diarrhea | 6
  Grade 3/4 Dehydration | 2
  Grade 5 Encephalopathy | 1
  Disease Progression NOS | 1

4. Secondary Outcome: Clinical Benefit Response Rate (Complete Response (CR)+Partial Response(PR)+Stable Disease(SD) > 180 Day Duration).
Time Frame: 18 months
Population: 20 evaluable subjects were analyzed for Clinical Benefit Rate (CR+PR+SD>180 days per RECIST criteria.
Measure: Number; unit: participants
Arm/Group | Lonafarnib
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: Duration of Study, a maximum of seven cycles (Typically 21 days)
Arm/Group | Lonafarnib
Serious Adverse Events (participants affected / at risk) | 7/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonafarnib (N=29)
ATAXIA (INCOORDINATION) (Nervous system disorders) | 1 (1)
DEATH NOT ASSOCIATED WITH CTCAE TERM / DISEASE PROGRESSION NOS (General disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 1 (2)
ENCEPHALOPATHY (Nervous system disorders) | 1 (2)
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
HEPATOBILIARY/PANCREAS - OTHER (Hepatobiliary disorders) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonafarnib (N=29)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 5 (7)
ALKALINE PHOSPHATASE (Investigations) | 5 (6)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 1 (1)
ALLERGY/IMMUNOLOGY - OTHER (Immune system disorders) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 3 (4)
ANOREXIA (Gastrointestinal disorders) | 17 (27)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 3 (3)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 8 (12)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (1)
BLOOD/BONE MARROW - OTHER (Blood and lymphatic system disorders) | 1 (1)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Investigations) | 1 (1)
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 2 (2)
CARDIAC GENERAL - OTHER (Cardiac disorders) | 1 (1)
CHELITIS (Skin and subcutaneous tissue disorders) | 1 (1)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 2 (2)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
COLITIS, INFECTIOUS (E.G., CLOSTRIDIUM DIFFICILE) (Gastrointestinal disorders) | 1 (1)
CONFUSION (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 15 (17)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (11)
CREATININE (Investigations) | 2 (6)
CYSTITIS (Renal and urinary disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 3 (3)
DERMAL CHANGE LYMPHEDEMA, PHLEBOLYMPHEDEMA (Blood and lymphatic system disorders) | 2 (2)
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 22 (57)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 6 (8)
DRY EYE SYNDROME (Eye disorders) | 2 (2)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 14 (16)
EDEMA: LIMB (Blood and lymphatic system disorders) | 2 (2)
EYELID DYSFUNCTION (Eye disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 25 (48)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (2)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
FLU-LIKE SYNDROME (General disorders) | 1 (1)
FLUSHING (Skin and subcutaneous tissue disorders) | 3 (3)
FRACTURE (Musculoskeletal and connective tissue disorders) | 2 (3)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 2 (3)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 3 (6)
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Investigations) | 2 (3)
GROWTH AND DEVELOPMENT - OTHER (General disorders) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 6 (6)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 6 (7)
HEMOGLOBIN (Blood and lymphatic system disorders) | 8 (10)
HOT FLASHES/FLUSHES (Endocrine disorders) | 9 (9)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (2)
HYPERTENSION (Cardiac disorders) | 3 (3)
INCONTINENCE, ANAL (Gastrointestinal disorders) | 1 (2)
INFECTIONWITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / SINUS (Infections and infestations) | 1 (1)
INFECTION - OTHER (Infections and infestations) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / WOUND (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 15 (18)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 2 (3)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 (5)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 10 (10)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 8 (8)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / STOMACH (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 4 (6)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 1 (3)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 18 (36)
NEUROLOGY - OTHER (Nervous system disorders) | 1 (1)
NEUROPATHY: MOTOR (Nervous system disorders) | 2 (2)
NEUROPATHY: SENSORY (Nervous system disorders) | 17 (17)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
OBESITY (General disorders) | 1 (1)
OBSTRUCTION/STENOSIS OF AIRWAY / BRONCHUS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OCULAR/VISUAL - OTHER (Eye disorders) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 5 (6)
PAIN / BACK (General disorders) | 8 (9)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN / BREAST (Reproductive system and breast disorders) | 1 (1)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 5 (5)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 7 (11)
PAIN / HEAD/HEADACHE (General disorders) | 6 (7)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 7 (13)
PAIN / NECK (General disorders) | 1 (1)
PAIN / PAIN NOS (General disorders) | 3 (5)
PAIN / PELVIS (General disorders) | 3 (4)
PAIN / STOMACH (Gastrointestinal disorders) | 1 (1)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / TUMOR PAIN (General disorders) | 1 (1)
PAIN - OTHER (General disorders) | 1 (1)
PANCREATIC ENDOCRINE: GLUCOSE INTOLERANCE (Endocrine disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 4 (4)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PORTAL VEIN FLOW (Vascular disorders) | 1 (1)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 4 (4)
PROLONGED QTC INTERVAL (Cardiac disorders) | 1 (2)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 7 (7)
PULMONARY FIBROSIS (RADIOGRAPHIC CHANGES) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 3 (3)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 3 (3)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (3)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 (1)
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 2 (2)
RIGORS/CHILLS (General disorders) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 5 (9)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 10 (12)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
THYROID FUNCTION, LOW (HYPOTHYROIDISM) (Endocrine disorders) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 13 (20)
WEIGHT GAIN (General disorders) | 1 (1)
WEIGHT LOSS (General disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No